CLINICAL TRIAL: NCT07175623
Title: Comparison of the Effects of the Interaction of Methylprednisolone and Dexamethasone With Sugammadex on Rocuronium Reversal Time, Postoperative Pain, and Nausea in Pediatric Patients: A Randomized Controlled Trial
Brief Title: Methylprednisolone vs Dexamethasone Interaction With Sugammadex in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, MUSTAFA BÜYÜKCAVLAK, Specialist in Anesthesiology and Intensive Care, Principal Investigator, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-5/2025
Record Dates: First submitted 2025-09-03; First posted 2025-09-16 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Neuromuscular Block, Residual; Pain Management; Postoperative Nausea
Keywords: Sugammadex; Methylprednisolone; Dexamethasone; Postoperative pain; Postoperative nausea; Pediatric Anesthesia
MeSH Terms: conditions — Delayed Emergence from Anesthesia; Agnosia; Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Methylprednisolone (Experimental): Patients will receive intravenous methylprednisolone 1 mg/kg at the induction of anesthesia.
  Interventions: Drug: Methyl Prednisolone (MP)
- Dexamethasone (Experimental): Patients will receive intravenous dexamethasone 0.2 mg/kg at the induction of anesthesia
  Interventions: Drug: Dexamethasone (0.2 mg/kg)
- Control (Placebo Comparator): Patients will receive 5 ml of intravenous normal saline at the induction of anesthesia
  Interventions: Drug: Saline (0.9% NaCl)

INTERVENTIONS:
Drug: Methyl Prednisolone (MP) — Dose: 1 mg/kg IV
  Timing: at the induction of anesthesia
  Arms: Methylprednisolone
Drug: Dexamethasone (0.2 mg/kg) — Dose: 0.2 mg/kg IV (glucocorticoid equivalent to 1 mg/kg methylprednisolone)
  Timing: at the induction of anesthesia
  Arms: Dexamethasone
Drug: Saline (0.9% NaCl) — Dose: 5 ml IV
  Timing: at the induction of anesthesia
  Arms: Control

SUMMARY:
This randomized controlled trial aims to compare the interaction of methylprednisolone and dexamethasone with sugammadex in pediatric patients undergoing adenoidectomy and/or tonsillectomy. The primary objective is to evaluate the effect of these corticosteroids on the reversal time of rocuronium-induced neuromuscular block by sugammadex. Secondary outcomes include postoperative pain, nausea and vomiting, extubation time, and adverse events. Eligible participants are children aged 5 to 12 years, ASA I-II, scheduled for elective surgery under general anesthesia. The study is designed as a triple-blind, parallel-group trial with three arms: methylprednisolone, dexamethasone, and placebo.

DETAILED DESCRIPTION:
Neuromuscular blocking agents (NMBAs) are widely used in pediatric anesthesia to facilitate tracheal intubation and optimize surgical conditions. However, residual neuromuscular block may increase the risk of postoperative respiratory complications, especially in children who have shorter safe apnea times due to their unique anatomical and physiological characteristics. Sugammadex, a modified γ-cyclodextrin, is a selective reversal agent for aminosteroid NMBAs such as rocuronium. Its mechanism of encapsulating steroidal neuromuscular blocking molecules raises concerns about potential interactions with other steroidal drugs, including perioperatively used corticosteroids.

Corticosteroids are commonly administered in the perioperative period for their antiemetic, analgesic, and anti-inflammatory effects. Dexamethasone is widely accepted for postoperative nausea and vomiting prophylaxis, while methylprednisolone is preferred for its rapid anti-inflammatory effect. Previous studies have suggested that the structural similarity of corticosteroids to rocuronium may interfere with sugammadex binding, but the available evidence is conflicting, and data on methylprednisolone remain limited. In a prior study, methylprednisolone was shown to prolong sugammadex reversal time slightly, but no direct comparison with another corticosteroid was performed.

This randomized controlled trial is designed to compare the effects of methylprednisolone and dexamethasone on sugammadex reversal time in pediatric patients undergoing adenoidectomy and/or tonsillectomy. The study will assess whether methylprednisolone has a stronger interaction with sugammadex compared with dexamethasone, leading to prolonged recovery from rocuronium block. Secondary outcomes will include postoperative pain, nausea and vomiting, extubation time, and adverse events. The results may provide clinically relevant evidence regarding the choice of corticosteroid in pediatric anesthesia when sugammadex is used for neuromuscular block reversal.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-12 years
* American Society of Anesthesiologists (ASA) physical status I-II

Exclusion Criteria:

* ASA physical status ≥ III
* Emergency surgery
* Known allergy or contraindication to neuromuscular blocking agents, sugammadex, or corticosteroids
* Chronic or recent systemic corticosteroid use (within the last 3 months)
* Neuromuscular disorders (e.g., muscular dystrophy, myasthenia gravis)
* Severe hepatic or renal dysfunction
* Significant respiratory or cardiac disease
* Anticipated difficult airway or history of difficult intubation
* Developmental delay or craniofacial anomalies affecting airway management
* Refusal of consent

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-09-16 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Time to recovery of neuromuscular function (normalised train-of-four ratio ≥ 0.9) after sugammadex injection | From intravenous administration of sugammadex until achievement of normalized TOF ratio ≥ 0.9 (in seconds).
  Time from intravenous sugammadex administration to restoration of normalised train-of-four ratio ≥ 0.9, measured by quantitative acceleromyography at the adductor pollicis muscle under standardized monitoring conditions.

SECONDARY OUTCOMES:
Extubation time | From intravenous administration of sugammadex until tracheal extubation (in minutes).
  Time from intravenous sugammadex administration to removal of the endotracheal tube, recorded by anesthesia staff.
Postoperative pain score | At 2 hours after surgery.
  Faces Pain Scale-Revised (0-10) assessed at predefined time points; higher scores indicate more pain.
Postoperative Nausea Severity | At 2 hours after surgery.
  Baxter Retching Faces (0-10) pictorial scale; higher scores indicate more severe nausea/retching.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Konya City Hospital, Konya, Karatay
  - Bezmialem Vakıf Univerisity Dragos Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gulec E, Biricik E, Turktan M, Hatipoglu Z, Unlugenc H. The Effect of Intravenous Dexamethasone on Sugammadex Reversal Time in Children Undergoing Adenotonsillectomy. Anesth Analg. 2016 Apr;122(4):1147-52. doi: 10.1213/ANE.0000000000001142. PMID 26771267
- [Background] Buonanno P, Laiola A, Palumbo C, Spinelli G, Servillo G, Di Minno RM, Cafiero T, Di Iorio C. Dexamethasone Does Not Inhibit Sugammadex Reversal After Rocuronium-Induced Neuromuscular Block. Anesth Analg. 2016 Jun;122(6):1826-30. doi: 10.1213/ANE.0000000000001294. PMID 27028777
- [Background] Murphy GS, Sherwani SS, Szokol JW, Avram MJ, Greenberg SB, Patel KM, Wade LD, Vaughn J, Gray J. Small-dose dexamethasone improves quality of recovery scores after elective cardiac surgery: a randomized, double-blind, placebo-controlled study. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):950-60. doi: 10.1053/j.jvca.2011.03.002. Epub 2011 May 11. PMID 21565530
- [Background] . Gold SJA, Harper NJN. The place of sugammadex in anaesthesia practice. Trends Anaesth Crit Care 2012; 2: 4-9.
- [Background] Graham LA, Illarmo S, Wren SM, Mudumbai SC, Odden MC. Optimal multimodal analgesia combinations to reduce pain and opioid use following non-cardiac surgery: an instrumental variable analysis. Reg Anesth Pain Med. 2025 Jul 17:rapm-2025-106720. doi: 10.1136/rapm-2025-106720. Online ahead of print. PMID 40659442
- [Background] Aouad MT, Nasr VG, Yazbeck-Karam VG, Bitar MA, Bou Khalil M, Beyrouthy O, Harfouche D, Terrin N, Siddik-Sayyid S. A comparison between dexamethasone and methylprednisolone for vomiting prophylaxis after tonsillectomy in inpatient children: a randomized trial. Anesth Analg. 2012 Oct;115(4):913-20. doi: 10.1213/ANE.0b013e3182652a6a. Epub 2012 Jul 13. PMID 22798534